CLINICAL TRIAL: NCT06189053
Title: Long-term Outcomes of Myocarditis Following Administration of SPIKEVAX (COVID-19 Vaccine mRNA)
Brief Title: A Study to Assess Long-term Outcomes of Myocarditis Following Administration of COVID-19 mRNA Vaccine (SPIKEVAX)
Status: Active, not recruiting | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mRNA-1273-P911
Record Dates: First submitted 2024-01-01; First posted 2024-01-03 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Myocarditis
Keywords: mRNA-1273; mRNA-1273 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — Myocarditis; Coronavirus Infections; Virus Diseases; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: Post-vaccine Myocarditis (PVM): Cohort 1 will include participants with a myocarditis event diagnosis or service date within 30 days on/after a SPIKEVAX vaccination and participants with at least 1 dose of SPIKEVAX in the 7 days prior to and including the index date.
- Cohort 2: All Other Myocarditis: Cohort 2 will include participants with no evidence of SPIKEVAX and no evidence of other vaccines targeting SARS CoV-2 within 30 days on/after a SPIKEVAX vaccination.

SUMMARY:
The main goal of this study is to characterize presentation, clinical course, and long-term outcomes of myocarditis temporally associated with administration of mRNA-1273 (SPIKEVAX) COVID-19 vaccine.

DETAILED DESCRIPTION:
This is an observational cohort study that combines data collected directly from healthcare providers (HCP) with existing retrospective real-world data as captured in clinical electronic health record (EHR) and administrative claims data. Vaccine exposure and case identification information will be obtained retrospectively from existing real-world data to identify cases of post-vaccine myocarditis (PVM) and ultimately vaccine-associated myocarditis (VAM) for potential study inclusion. Eligible participants will be identified and followed for up to 5 years until the end of the study period or loss to follow-up or death.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of myocarditis between December 18, 2020, and October 31, 2026, will be identified or who have a relevant combination of laboratory and clinical findings meeting the CDC case definition for probable or confirmed myocarditis will be included in the study.
* Participants will be required to have at least 30 days of medical history to assess SPIKEVAX exposure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The source population for this study will include participants with a diagnosis of myocarditis or a relevant combination of laboratory and clinical findings meeting the Centers for Disease Control and Prevention (CDC) case definition for probable or confirmed myocarditis occurring during the study window for case ascertainment.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Major Adverse Clinical Outcomes | Up to 5 years
  Adverse clinical outcomes may include myocardial infarction, heart failure, stroke, and cardiovascular hospitalization.
Number of Participants with Persistent Cardiac Abnormality | Up to 5 years
Functional Assessment: Number of Participants Reporting Symptoms of Chest Pain, Dyspnea, Palpitations, and Syncope | Up to 5 years
Functional Assessment: Number of Participants Returning to Normal Activities | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Veradigm, Chicago, Illinois, United States